CLINICAL TRIAL: NCT00596310
Title: Early Detection of Lung Cancer in a High-Risk Population Defined by Pulmonary Function Testing, Biomarkers, and Computerized Tomography Scanning
Brief Title: Early Detection of Lung Cancer in a High-Risk Population Defined by PFT, Biomarkers, and CT Scanning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Susanne Arnold (Other)
Collaborators: Marty Driesler Cancer Project (Unknown); Kentucky Lung Cancer Research Program (Other)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Associate Director for Clinical Translation, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MDCP-Lung
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer; screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Screening CT
  Interventions: Other: CT

INTERVENTIONS:
Other: CT — Screening CT

SUMMARY:
Lung cancer is the number one cancer killer in Kentucky and has a very high incidence within the 5th Congressional District of Kentucky (110.8 cases per 100,000 in period 1996-2000). Surgical removal provides the best chance for cure. Unfortunately, the majority of lung cancer cases are detected in an advanced stage, when surgical resection is impossible. This leads to shorter survival rates and increased mortality rates for lung cancer, increased patient suffering, and greater cost to the healthcare system. Methods that favor earlier detection are therefore crucial for successful treatment. One such method, low-dose spiral computed tomography (CT) is being studied to determine whether its use as a screening method will lead to earlier detection and earlier intervention, perhaps impacting survival and mortality in lung cancer. This method has a modest sensitivity to detect lung cancer, but low specificity, which leads to many false positives and a low negative predictive value. The present study is designed to address both of these limitations by: 1) identifying individuals in the population at highest risk for developing lung cancer (due to smoking habits and decreased pulmonary function) for subsequent CT screening, and 2) performing biomarker testing in conjunction with the CT scan to improve the ability to discern individuals with benign lung nodules from those with malignant tumors. The 5th Congressional District of Kentucky has one of the highest rates of lung cancer in the nation and is an ideal location to test the validity (sensitivity and specificity), feasibility (negative and positive predictive value), and efficacy (stage distribution shift to earlier stage disease, increased survival, and decreased cancer-specific mortality) of these strategies to enhance early detection.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-75 years old.
* Identification of a primary care physician (can be identified by study staff if needed).
* FEV1/FVC <70% (GOLD 1 or higher COPD) (poor breathing function).
* > or = 40 pack-year current or former (within the last 10 years) tobacco use (i.e. heavy cigarette smoking history).

Exclusion Criteria:

* Enrolled in any other lung screening or lung cancer prevention trial.
* Chest CT within the prior 12 months.
* Inability to lie flat with arms raised above the head.
* Current or prior personal history of lung cancer.
* Prior history of cancer within the last five years or currently receiving treatment for cancer, except adequately treated non-melanomatous skin cancer or in-situ cervical cancer.
* Life expectancy of less than 5 years.
* Patients requiring supplemental oxygen.
* Inability to give informed consent.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
test validity | 5 years

SECONDARY OUTCOMES:
test feasibility | 5 years
test efficacy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Arnold, M.D., Principal Investigator — University of Kentucky
Locations (4):
- United States (4):
  - Hazard ARH Regional Medical Center, Hazard, Kentucky
  - St. Claire Regional Medical Center, Morehead, Kentucky
  - Highlands Regional Medical Center, Prestonsburg, Kentucky
  - Lake Cumberland Regional Hospital, Somerset, Kentucky

IPD SHARING:
Plan to Share IPD: No